CLINICAL TRIAL: NCT06820775
Title: EFFECTIVENESS OF A TRIPLE NUTRITIONAL INTERVENTION AND PHYSICAL ACTIVITY FOR GLYCOSYLATED HB CONTROL IN PREDIABETICS: CLINICAL TRIAL
Brief Title: EFFECTIVENESS OF A TRIPLE NUTRITIONAL INTERVENTION AND PHYSICAL IN PREDIABETIC PATIENRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioaraba Health Research Institute (Network)
Responsible Party: Principal Investigator, ANTXON APIÑANIZ, GENERAL PRACTITIONNER, Osakidetza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREDIABET01
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Diabetes
Keywords: DIABETES MELLITUS
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTIONAL GROUP (Experimental): Health advice and triple intervention: 15 ml apple cider vinegar diluted in a glass of water before meals, order in the sequence of meals (sequence of food intake: first vegetables, second proteins, third fats and finally carbohydrates) and physical activity immediately after meals.
  Description of all interventions:
  Patients in both groups: all patients will receive health advice on sports practice from the WHO, Osakidetza and the Basque Government (42-44).
  Likewise, the nurse will give healthy eating recommendations according to the Osakidetza guide (41):
  1.1 Recommendation sports practice: ecommendation 1:
  >>All persons aged 18 years and older should accumulate a minimum of 150 minutes per week of moderate aerobic physical activity, or 75 minutes of vigorous aerobic physical activity each week, or an equivalent combination of moderate and vigorous activities. Exercise should be in sessions of at least 10 minutes.
  Recommendation 2: Twice or more times per week, it is advisable to
  Interventions: Combination Product: A TRIPLE INTERVENTION NUTRITION AND PHYSICAL ACTIVITY
- CONTROL GROUP (No Intervention): Patients will receive the same attention as provided in routine clinical practice,

INTERVENTIONS:
Combination Product: A TRIPLE INTERVENTION NUTRITION AND PHYSICAL ACTIVITY — Intervention group: Health advice and triple intervention: 15 ml apple cider vinegar diluted in a glass of water before meals, order in the sequence of meals (sequence of food intake: first vegetables, second proteins, third fats and finally carbohydrates) and physical activity immediately after meals.
  Description of all interventions:
  Patients in both groups: all patients will receive health advice on sports practice from the WHO, Osakidetza and the Basque Government.
  Arms: INTERVENTIONAL GROUP

SUMMARY:
Diabetes represents a substantial burden on health care systems. People with prediabetes IGT (impaired glucose tolerance) or IFG (impaired fasting glucose) are at high risk of developing diabetes, and up to 50% progress to diabetes within 5 years.

OBJECTIVE: To evaluate the effectiveness of a triple intervention (physical activity and ordered healthy diet) to improve glycosylated hemoglobin control in prediabetic patients.

MATERIAL AND METHODOLOGY: Randomized, open, controlled clinical trial with routine clinical practice (health advice for physical activity and healthy diet). Study population: obese or overweight patients of the OSI Araba aged 35-70 years who are in the contemplation stage.

Response assessment: Primary variable: glycosylated hemoglobin; Secondary variables: Body Mass Index (BMI) (kg/cm2); blood pressure (mm Hg); satisfaction questionnaire score; physical exercise index (IPAQ) (METs). Statistical analysis: The analysis of the main variable (change in HbA1c at 6 months between both groups) will be assessed by analysis of covariance, ANCOVA, adjusting for baseline HbA1c. Sample size: 41 patients per arm (+30% to cover losses to follow-up).

ELIGIBILITY:
Inclusion Criteria:

Prediabetics with glycosylated hemoglobin (HbA1c) 5.7-6.4 (24, 38) and signing informed consent.

-

Exclusion Criteria:

Presence of physical or psychological illnesses that prevent physical activity; participation in another research project; pregnancy or breastfeeding; patients undergoing dietary or pharmacological treatment for weight loss; history of myocardial infarction or stroke; diabetic, taking drugs for diabetes mellitus and taking drugs such as Gliflozin for pathologies other than diabetes mellitus.

of physical or psychological illnesses that prevent physical activity; participation in another research project; pregnancy or breastfeeding; patients undergoing dietary or pharmacological treatment for weight loss; history of myocardial infarction or stroke; diabetic, taking drugs for diabetes mellitus and taking drugs such as Gliflozin for pathologies other than diabetes mellitus.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-02-02 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | At baseline, 3 and 6 months
  Glycated hemoglobin (HbA1c)

SECONDARY OUTCOMES:
BMI (kg/cm2) | At baseline, 3 and 6 months
  BMI (kg/cm2)
Satisfaction of patients | At 6 months
  Score in the satisfaction questionnaire
Physical exercise index | At baseline, 3 and 6 months
  Physical exercise index (IPAQ)
Compliance with the triple dietary intervention | At 3 and 6 months
  Compliance with the triple dietary intervention
Percentage of patients who reach normoglycemia (HbA1c < 5.7) | At 3 and 6 months
  Prcentage of patients who reach normoglycemia (HbA1c < 5.7).

CONTACTS AND LOCATIONS:
Locations (1):
- Antxon Apiñaniz, Vitoria-Gasteiz, Alava, Spain